CLINICAL TRIAL: NCT05665894
Title: Vacuum-Assisted Evacuation (VAE) Of Symptomatic and/or Voluminous Breast Haematomas Following Surgeries And Percutaneous Procedures: a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Marco Materazzo, Phd Student, University of Rome Tor Vergata
Other Study IDs: BREAST HEMATOMA
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Breast Haematoma; Breast Cancer; Breast Diseases
Keywords: Breast Neoplasm; Breast Hematoma; Breast Diseases; Vaacum assisted biopsy
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Breast hematoma group: Patients of age between 18 and 75 years old after breast conservative surgery (BCS), VAB or vacuum-assisted excision (VAE) procedure in our facility, who developed clinically significant and large hematoma (>25 mm). In our institution, we routinely offer a trial of Vacuum-Assisted Evacuation (VAEv) for >25 mm hematoma that does not fulfill the criteria for immediate surgery and causes discomfort, pressure symptoms, infection, or pain classified on VAS > 3.
  Interventions: Device: Hematoma Vaacum Assisted Biopsy

INTERVENTIONS:
Device: Hematoma Vaacum Assisted Biopsy — The patient was placed supine and meticulous aseptic measures were applied. Prior procedure local anesthesia (lidocaine 1%) was administered following disinfection. A 5 mm skin incision is performed to guarantee appropriate access for the needle insertion in the hematomas. The evacuation was achieved using a Mammotome® vacuum-assisted system (Devicor Medical Products, Inc., Cincinnati, OH, USA), with an 8-G needle, under the guidance of the same high-resolution US equipment (MyLabTM 9 XP; Esaote SpA, Genoa) for preoperative assessment. Empty-needle function and the tissue-biopsy option is preferred to fragment the fibrotic tissue until the hematoma empties and its walls collapsed. Once VAEv is performed, the postoperative US is carried out and VAEv is repeated until more than 90% evacuations of hematoma volume if no complication occurs.
  Other Names: Hematoma Core needle biopsy

SUMMARY:
Among postoperative complications in breast surgery, hematoma is the most common occurrence. While mostly self-limited, in some cases surgical revision is mandatory when hematoma occurs. Among percutaneous procedures, preliminary studies demonstrated the efficacy of vacuum-assisted breast biopsy(VAB) in evacuating breast hematomas. The aim of the present study is to investigate the efficacy of VAB system in evacuating hematoma, symptoms resolution, and avoidance of surgery.

From January 2016 to January 2020 ≥25 mm symptomatic breast hematoma after breast conserving surgery(BCS) and percutaneous procedures were retrospectively enrolled from a perspective maintained database. Preoperative demographic and clinical data were collected. Hematoma maximum diameter, Estimated hematoma volume, total procedure time, and visual analog scale (VAS) score prior ultrasound(US) Vacuum-Assisted Evacuation (VAEv) were recorded. At one week VAS score, residual hematoma volume, and complications were recorded. Study outcomes were defined as clearance of ≥70% postoperative hematoma, symptoms resolution (assessed as patient report visual analog scale (VAS≤3)), and avoidance of surgery during follow-up.

DETAILED DESCRIPTION:
A monocentric, retrospective study from a prospectively maintained database was planned to evaluate the clinical outcome of patients undergoing VAB procedures for postoperative breast hematoma between 1st January 2016 and 1st January 2020.

Once breast hematoma is diagnosed and FNA did not obtain a complete clearance of the hematoma, in our clinical practice VAEv procedure is planned between 10-14 days from the first procedure (surgery, VAB, VAE). All VAEv procedures are performed in our outpatient department by a radiologist with > 10 years of experience in breast imaging and US-guided procedures.

Preoperative assessment is carried out just prior VAEv with high-resolution ultrasound (US) equipment (MyLabTM 9 XP; Esaote SpA, Genoa, Italy) and with 10-13 MHz linear array transducer (Esaote SpA, Genoa, Italy). The patient was placed supine and meticulous aseptic measures were applied. Prior procedure local anesthesia (lidocaine 1%) was administered following disinfection. A 5 mm skin incision is performed to guarantee appropriate access for the needle insertion in the hematomas. The evacuation was achieved using a Mammotome® vacuum-assisted system (Devicor Medical Products, Inc., Cincinnati, OH, USA), with an 8-G needle, under the guidance of the same high-resolution US equipment (MyLabTM 9 XP; Esaote SpA, Genoa) for preoperative assessment. Empty-needle function and the tissue-biopsy option is preferred to fragment the fibrotic tissue until the hematoma empties and its walls collapsed. Once VAEv is performed, the postoperative US is carried out and VAEv is repeated until more than 90% evacuations of hematoma volume if no complication occurs.

If the hematoma occurred after the percutaneous procedure (VAB, VAE), a new metal clip is placed in the site of the procedure to locate target breast lesion. At the end of the procedure, the hematoma site is then manually compressed for 5-10 min. Finally, the surgical site is covered with dressings and locoregional ice therapy was applied. Usually, after VAEv patients were observed in our outpatient clinic for 3 hours after the procedure prior to home discharge.

All patients were advised to wear tight sports-brassiere was recommended for a minimum of 24 hours to prevent rebleeding or major seroma formation. After VAEv patients are educated regarding our telephonic follow-up for any symptoms onset and are routinely re-evaluated at 1 week with US examination (MyLabTM 9 XP; Esaote SpA, Genoa, Italy) with 10-13 MHz linear array transducer (Esaote SpA, Genoa, Italy), VAS assessment, and postoperative complications. Further telephonic follow-up evaluation is routinely scheduled to avoid late symptomatic breast hematoma underestimation.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years old after breast conservative surgery (BCS), VAB or vacuum-assisted excision (VAE) procedure
* Clinically significant and large hematoma (>25 mm) that do not fulfill the criteria for immediate surgery and cause discomfort, pressure symptoms, infection, or pain classified on VAS > 3.
* Failure of attempt with FNA
* Patients that refuse surgery

Exclusion Criteria:

* pregnancy
* patients requiring urgent surgery
* Patient follow-up discontinued in our facility
* Symptomatic post-BCS early hematoma

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Study Population: All female patients that developed postoperative or postoprocedural breast hematoma which do not requires urgent surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Hematoma vacuum assisted biopsy success rate I | At the end of the procedure
  Clearance of ≥70% postoperative hematoma
Symptom Resolution | At the end of the procedure
  Patient report visual analog scale (VAS) ≤3 (minimum 0; maximum 10) at the end of Hematoma vacuum assisted biopsy
Hematoma vacuum assisted biopsy success rate I | 30 days from the procedure
  Avoidance of surgery during follow-up for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Tor Vergata University Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almasarweh S, Sudah M, Joukainen S, Okuma H, Vanninen R, Masarwah A. The feasibility of ultrasound-guided vacuum-assisted evacuation of large breast hematomas. Radiol Oncol. 2020 Jun 26;54(3):311-316. doi: 10.2478/raon-2020-0041. PMID 32598321
- [Background] Guzman-Aroca F, Berna-Serna JD, Garcia-Ortega AA, Hernandez-Gomez D, Berna-Mestre JD. A New Management Technique for Symptomatic Haematomas Following Therapeutic Vacuum-Assisted Biopsy. J Clin Med. 2019 Sep 19;8(9):1493. doi: 10.3390/jcm8091493. PMID 31546843